CLINICAL TRIAL: NCT06995274
Title: Umbilical Cord Blood Therapy in a Child With Eosinophilic Duodenitis and Autism Spectrum Disorder: a Case Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principle Investigator, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-03-057
Record Dates: First submitted 2025-05-11; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Eosinophilic Gastrointestinal Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- umbilical cord blood (Experimental): This is a single-arm, open-label, exploratory case study involving one pediatric participant diagnosed with both eosinophilic duodenitis (ED) and autism spectrum disorder (ASD). The intervention includes a series of three intravenous umbilical cord blood (UCB) infusions: one autologous UCB infusion followed by two allogeneic UCB infusions at 6-week intervals. Each infusion is performed under sterile conditions at a hospital-based cell therapy center. The donor UCB units are selected based on HLA compatibility (minimum 3/6 match for HLA-A, B, DRB1) and total nucleated cell count (≥ 3×10⁷ cells/kg). The allogeneic infusions are accompanied by a 7-day low-dose oral cyclosporine regimen to reduce the risk of immune rejection. The total study period includes baseline evaluation, three infusion sessions, and multiple post-infusion follow-up assessments over three months.
  Interventions: Biological: Umbilical Cord Blood Infusion (Autologous and Allogeneic)

INTERVENTIONS:
Biological: Umbilical Cord Blood Infusion (Autologous and Allogeneic) — The intervention consists of three intravenous infusions of umbilical cord blood (UCB) in a pediatric patient diagnosed with both eosinophilic duodenitis (ED) and autism spectrum disorder (ASD). The first infusion uses autologous UCB stored at a certified cord blood bank. The second and third infusions use allogeneic UCB units selected from a hospital-based donor cord blood bank. Donor units are matched at a minimum of 3 out of 6 HLA loci (HLA-A, B, DRB1) and contain ≥ 3×10⁷ total nucleated cells per kilogram of body weight.
  Each infusion is administered intravenously via peripheral vein at the Cell Therapy Center of CHA Bundang Medical Center. Prior to each infusion, the participant receives premedication with intravenous chlorpheniramine maleate (0.6 mL/10 kg) to reduce the risk of allergic reactions. For allogeneic infusions, oral cyclosporine (0.07 mL/kg twice daily) is administered for 7 days (3 days before, day of, and 3 days after infusion) to minimize immune-mediated reactions

SUMMARY:
This single-case exploratory clinical study aims to evaluate the therapeutic potential of umbilical cord blood (UCB) infusion in a pediatric patient diagnosed with both eosinophilic duodenitis (ED) and autism spectrum disorder (ASD). ED is a rare inflammatory gastrointestinal condition characterized by excessive eosinophil infiltration in the duodenal mucosa, often associated with immune hypersensitivity and allergic responses. ASD is a neurodevelopmental disorder marked by deficits in social interaction, communication, and behavioral flexibility. Recent evidence suggests a link between gastrointestinal inflammation and neurodevelopmental symptoms via the gut-brain axis, especially in patients with co-occurring ASD and eosinophilic gastrointestinal disorders (EGIDs).

In this study, the patient will receive three UCB infusions: one autologous and two allogeneic. The first (autologous) UCB is stored at a certified cord blood bank and will be administered intravenously. Subsequently, two allogeneic UCB infusions will be administered six weeks apart using HLA-matched donor units selected from a hospital-based cord blood repository. The cell product will contain a minimum of 3 × 10⁷ total nucleated cells per kg, and donor-recipient compatibility for HLA A, B, and DRB1 will be considered.

To support immune tolerance and reduce potential adverse responses, a 7-day course of low-dose oral cyclosporine will be administered with each allogeneic infusion. All cord blood handling, thawing, and infusion will be performed in a cell therapy center under standardized protocols.

The primary aim is to explore the immune regulatory effects and symptom relief following UCB therapy in this rare comorbid case. Assessments will include brain MRI with DTI, EEG, fNIRS, sensory profiles (SP), social communication questionnaires (SCQ), autism rating scales (K-CARS-2), behavioral checklists (CBCL), gastrointestinal endoscopy, and developmental/cognitive/language assessments (e.g., WISC, WPPSI, GMFM, VMI, SELSI, PRES, FIM). Blood samples will be analyzed for eosinophil counts and gene/protein expression related to inflammation, neuroendocrine function, and gut-brain signaling (e.g., TNF-α, IL-6, serotonin, dopamine, GABA, CRH, BDNF).

This case study will also track safety indicators including vital signs, laboratory panels, and adverse events. The data may inform the feasibility of future therapeutic use of UCB in children with complex immune-neurodevelopmental conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Child aged 4 years at the time of enrollment
2. Diagnosed with both eosinophilic duodenitis (ED) and autism spectrum disorder (ASD)
3. Actively receiving outpatient care at the Department of Rehabilitation Medicine, CHA Bundang Medical Center
4. Autologous cord blood available and stored at an accredited cord blood bank
5. Written informed consent provided by a legally authorized representative (parent or guardian) after receiving a full explanation of the study

Exclusion Criteria:

1. Presence of a severe uncontrolled medical condition that may interfere with cord blood infusion or study assessments
2. History of severe allergic reaction to components of the investigational product or immunosuppressive agents (e.g., cyclosporine)
3. Current or recent participation (within 30 days) in another interventional clinical trial
4. Any contraindication to MRI, EEG, or fNIRS assessments (e.g., implanted metal device, severe behavioral intolerance)
5. Determined by the principal investigator to be unsuitable for participation due to safety concerns or noncompliance

Ages: 4 Years to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Safety of Umbilical Cord Blood Infusion in a Child with Eosinophilic Duodenitis and Autism Spectrum Disorder | From baseline (within 6 months prior to first infusion) through 3 months after the final (third) UCB infusion (approximately 4-5 months total)
  The number and severity of adverse events (AEs) and serious adverse events (SAEs) related to cord blood infusion will be assessed and categorized using MedDRA and CTCAE v5.0. Unit of measure is number of participants with AE or SAE

SECONDARY OUTCOMES:
Change in Sensory Processing Scores (Sensory Profile) | Baseline (within 6 months prior to first infusion), 7 days after each infusion, and 3 months after final infusion
  To evaluate changes in sensory processing characteristics following umbilical cord blood (UCB) therapy using the Sensory Profile (SP), a standardized parent-report questionnaire assessing how sensory processing affects daily functioning. Improvement may indicate reduced sensory dysregulation, a common feature in ASD.
Change in Social Communication (SCQ Score) | Baseline, 7 days after each infusion, and 3 months after final infusion
  To assess changes in social communication behaviors and core ASD symptoms using the Social Communication Questionnaire (SCQ). These tools measure social reciprocity, communication, and autism symptom severity. Unit of Measure: Points (0-40)
Change in Behavioral Functioning (CBCL) | Baseline, 7 days after each infusion, and 3 months after final infusion
  To monitor changes in behavioral and emotional functioning using the Child Behavior Checklist (CBCL), a standardized parent-report measure of internalizing and externalizing behaviors. Unit of Measure: Points
Change in Brain Connectivity and White Matter Integrity (MRI with DTI) | Baseline and 3 months after final infusion
  Measures white matter integrity via fractional anisotropy from DTI scans.Unit of Measure: FA value (unitless, 0-1 scale)
Change in Cortical Hemodynamic Response (fNIRS) | Baseline and 3 months after final infusion
  To assess changes in prefrontal cortex activation during social and cognitive tasks using functional near-infrared spectroscopy (fNIRS), particularly during facial expression recognition and resting-state conditions. Unit of Measure: μmol/L
Change in EEG Patterns | Baseline and 3 months after final infusion
  EEG analysis of relative power in frequency bands, pre-post UCB herapy, using AI (iSyncBrain).Unit of Measure: μV²/Hz
Duodenal Eosinophil Count (if clinically indicated) | Baseline, 7 days after each infusion, and 3 months after final infusion
  Duodenal Eosinophil Count (if clinically indicated) Unit of Measure: Eosinophils per high power field (HPF)
Change in Autism Severity (K-CARS-2) | Baseline, 7 days after each infusion, and 3 months after final infusion
  To assess changes in core ASD symptoms using the Korean-Childhood Autism Rating Scale, 2nd Edition (K-CARS-2). These tools measure social reciprocity, communication, and autism symptom severity. Unit of Measure: Points (15-60)
Peripheral Blood Eosinophil Count | Baseline, 7 days after each infusion, and 3 months after final infusion
  Change in Gastrointestinal Inflammation, Cells/μL

IPD SHARING:
Plan to Share IPD: No